CLINICAL TRIAL: NCT02083055
Title: Anesthetic Advantages of Dexmedetomidine Compared With Nitroglycerin for Hypotensive Anesthesia in Orthognathic Surgery. A Randomized Clinical Trial.
Brief Title: Anesthetic Advantages of Dexmedetomidine for Hypotensive Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Duangdee Rummasak, department of oral and maxillofacial surgery, faculty of dentistry, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-DT/PY-IRB 2012/021.1904
Record Dates: First submitted 2014-03-06; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Anesthesia; Hypotension
Keywords: dexmedetomidine; controlled hypotensive anesthesia
MeSH Terms: conditions — Hypotension | interventions — Dexmedetomidine; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Experimental): Intraoperative controlled hypotension by dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- nitroglycerin (Active Comparator): Intraoperative controlled hypotension by nitroglycerin
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Dexmedetomidine — controlled hypotensive anesthesia with dexmedetomidine compare with nitroglycerin on anesthetic outcome such as analgesic use, time to eye opening, follow verbal command, extubation and early postoperative pain
  Other Names: precedex
  Arms: dexmedetomidine
Drug: Nitroglycerin — controlled hypotensive anesthesia with nitroglycerin compared with dexmedetomidine on anesthetic outcomes such as analgesic use, time to eye opening, follow verbal command, extubation, and early postoperative pain.
  Other Names: nitrocine
  Arms: nitroglycerin

SUMMARY:
The aim of this study was to evaluate the positive anesthetic properties such as reduce intraoperative analgesic requirement, time to extubation and recovery, and early postoperative pain of dexmedetomidine used as a hypotensive agent compared with nitroglycerin.

DETAILED DESCRIPTION:
The subject included the healthy patients who underwent orthognathic surgery and gave written the informed consent. The sample size was calculate from the amount of fentanyl use in orthognathic surgical case and difference more 30% was significant. Randomization was done by random number table to 2 groups. Both groups received standardized controlled hypotensive anesthesia and surgery. D group used dexmedetomidine as the hypotensive drug and N group use nitroglycerin. The main outcome were the amount of fentanyl use, time to eye opening, follow simple command, extubation, early postoperative pain, and early postoperative amount of pain killer. All recorded by anesthesiologist on data sheet.

compare statistical analysis used compare mean by unpaired student t test.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo bimaxillary surgery physical status I according to the classification of the American Society of Anesthesiologist age 18-45 years

Exclusion Criteria:

* systemic diseases not given informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
amount of intraoperative fentanyl | intraoperatve period
  Record the amount of fentanyl used in the operation.

SECONDARY OUTCOMES:
time to eye opening | emergence of anesthesia
  the time that counted from closed anesthetic drugs and reversed muscle relaxant to patients eye opening.
time to follow verbal command | emergence of anesthesia
  the time that counted from closed anesthetic drugs and reversed muscle relaxant to patients can follow simple verbal command such as open mouth, protrude the tongue, move the hand.
time to extubation | emergence of anesthesia
  the time that counted from closed anesthetic drugs and reversed muscle relaxant to remove the nasotracheal tube.
postoperative pain score at 30 minute | early postoperative period
  postoperative pain score at 30 minute using 10-point pain assessment scale.
postoperative pain score at 60 minute | early postoperative period
  postoperative pain score at 60 minute using 10-point pain assessment scale.
amount of pethidine | early postoperative period (first 2 hours)
  Record the amount of pethidine that used for a pain killer when pain score more than 4 in first 2 hours post-operation.

CONTACTS AND LOCATIONS:
Overall Officials: Duangdee Rummasak, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of dentistry, Mahidol university, Rajthevi, Bangkok, Thailand

REFERENCES:
- [Background] Apipan B, Rummasak D. Efficacy and safety of oral propranolol premedication to reduce reflex tachycardia during hypotensive anesthesia with sodium nitroprusside in orthognathic surgery: a double-blind randomized clinical trial. J Oral Maxillofac Surg. 2010 Jan;68(1):120-4. doi: 10.1016/j.joms.2009.07.065. PMID 20006165
- [Background] Rummasak D, Apipan B, Kaewpradup P. Factors that determine intraoperative blood loss in bimaxillary osteotomies and the need for preoperative blood preparation. J Oral Maxillofac Surg. 2011 Nov;69(11):e456-60. doi: 10.1016/j.joms.2011.02.085. Epub 2011 Jul 2. PMID 21724315
- [Background] Pineiro-Aguilar A, Somoza-Martin M, Gandara-Rey JM, Garcia-Garcia A. Blood loss in orthognathic surgery: a systematic review. J Oral Maxillofac Surg. 2011 Mar;69(3):885-92. doi: 10.1016/j.joms.2010.07.019. Epub 2010 Dec 31. PMID 21195531
- [Background] Choi WS, Samman N. Risks and benefits of deliberate hypotension in anaesthesia: a systematic review. Int J Oral Maxillofac Surg. 2008 Aug;37(8):687-703. doi: 10.1016/j.ijom.2008.03.011. Epub 2008 Jun 3. PMID 18511238
- [Background] Praveen K, Narayanan V, Muthusekhar MR, Baig MF. Hypotensive anaesthesia and blood loss in orthognathic surgery: a clinical study. Br J Oral Maxillofac Surg. 2001 Apr;39(2):138-40. doi: 10.1054/bjom.2000.0593. PMID 11286449
- [Background] El-Gohary MM, Arafa AS. Dexmedetomidine as ahypotensive agent: efficacy and hemodynamic response during spinal surgery for idiopathic scoliosis in adolescents. Egyptain Journal of Aanesthesia 2010; 26: 305-11.